CLINICAL TRIAL: NCT06013943
Title: Envafolimab Combined With GEMOX in First-line Treatment of Advanced Gallbladder Cancer : A Single Center, Single Arm, Phase II Trial
Brief Title: Envafolimab Combined With GEMOX in First-line Treatment of Advanced GBC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, Shen Feng, Professor and Chief Surgeon, Eastern Hepatobiliary Surgery Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EHBHKY2022-H040-P001
Record Dates: First submitted 2023-04-12; First posted 2023-08-28 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Gallbladder Cancer
Keywords: Envafolimab(immune checkpoint inhibitor anti-PD-L1 antibody)
MeSH Terms: conditions — Gallbladder Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Envafolimab+Gemox (Experimental)
  Interventions: Drug: Envafolimab+Gemox

INTERVENTIONS:
Drug: Envafolimab+Gemox — All of drugs were used for 6-8 cycles at the combined treatment stage, then Envafolimab and Gemcitabine continued at maintenance treatment stage until disease progression as defined by RECIST1.1, unacceptable toxicity, withdrawal from the study or death, or no more than 1 years.
  Combined treatment stage: Envafolimab(150mg, iH, Q1W, Day1)+Gemcitabine(1000mg/m2, iv, Q3W, Day1 and Day8)+Cisplatin(1000mg/m2, iv, Q3W, Day1 and Day8);
  Caintenance treatment stage: Envafolimab(400mg, iH, Day1, Q3W)+Gemcitabine(1000mg/m2, po, Day1-14, Q3W).

SUMMARY:
The TOPAZ-1 study compared the advantages and disadvantages of immune checkpoint inhibitor anti-PD-L1 antibody combined with Gem/Cis chemotherapy (Gemcitabine and Cisplatin) and Gem/Cis chemotherapy alone in first-line treatment of advanced biliary tract tumors (BTC, which including gallbladder cancer). It was observed that chemotherapy combined with PD-L1 antibody improved progression-free survival (PFS) and overall survival (OS).

As a standard first-line chemotherapy regimen for BTC too, Gemox chemotherapy (gemcitabine and cisplatin) has a median OS of 9.5 months, and non-inferior survival time to Gem/Cis chemotherapy. In addition, Gemox chemotherapy has been widely used in clinical practice because it reduces the requirement on patients' renal function and has good tolerance. Envafolimab is a novel fusion of humanized mono-domain PD-L1 antibody and human IgG Fc fragment, which has shown good efficacy and safety in a variety of solid tumors. It is safe and convenient to administer by subcutaneous injection. However, there is currently no clinical data on Envafolimab combined with GEMOX chemotherapy in patients with advanced gallbladder cancer (GBC).

The goal of this clinical trial is to evaluate its efficacy and related safety in patients with GBC. Eligible participants will receive Envafolimab (up to 12 months) plus gemcitabine and cisplatin (up to 6-8 cycles) until progression of radiological disease, unacceptable toxicity, or withdrawal from the study, whichever comes first.The primary endpoint was the 6-month PFS rate.

ELIGIBILITY:
Inclusion Criteria:

1. Definite diagnosis of gallbladder carcinoma by histology or cytology；
2. There is at least one measurable lesion (according to RECIST1.1);
3. From 18 to 75 years old, ECOG physical strength score of 0-2;
4. Basically normal bone marrow function: neutrophils >1.5x10^9/L, platelets >100x10^9/L;
5. Adequate renal function: creatinine clearance > 60ml/min;
6. Adequate liver function: bilirubin ≤1.5ULN;
7. No cardiac insufficiency or chest pain (medically uncontrollable); No myocardial infarction in the 12 months prior to study initiation;
8. Estimated survival time ≥3 months;
9. The patient must sign an informed consent form.

Exclusion Criteria:

1. Previous systematic therapy, including chemotherapy, immunotherapy and targeted therapy;
2. Secondary malignancies or other neoplasms (except superficial skin cancer and localized low-grade malignancies) occurring in the 3 years prior to study initiation;
3. The presence of brain or meningeal metastasis;
4. Have active or previously recorded autoimmune or inflammatory diseases (eg Rheumatoid arthritis, psoriasis, systemic lupus erythematosus, AIDS, etc. );
5. Have received allogeneic organ transplantation (eg kidney transplantation, liver transplantation, heart transplantation, etc. );
6. Patients who need long-term oral hormone therapy due to their underlying diseases;
7. Patients with interstitial pneumonia and autoimmune hepatitis;
8. Inflammatory infections during the active period of infection or other patients who may have disabilities receive planned treatment;
9. Persons with a history of uncontrolled substance abuse or mental disorders;
10. Patients with concomitant diseases that, in the judgment of the investigator, may seriously endanger their own safety or may interfere with the completion of the study;
11. Patients with poor renal function;
12. Untreated complete/incomplete ileus that prevents eating or interferes with systemic administration;
13. Participated in other clinical trials;
14. Pregnant and lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
6-month progression-free survival rate (PFS) | 6 months
  Defined as the rate of patients had no disease progression or death (whichever occurred first) from the start of treatment to 6 months after treatment.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to two years
  Defined as the time from the start of treatment to the date of progressive disease, or death, whichever occurred first.
Overall survival (OS) | Up to two years
  Defined as the time from the start of treatment to the date of death from any cause.
Disease control rate (DCR) per RECIST 1.1 | Once every 3 weeks (±7 days) from the first day of Envafolimab treatment for a maximum of 2 years until confirmed objective disease progression, death, and study termination.
  Defined as patients achieving a complete response [CR] or partial response [PR] or stable disease [SD].
Objective response rate (ORR) per RECIST 1.1 | Once every 3 weeks (±7 days) from the first day of Envafolimab treatment for a maximum of 2 years until confirmed objective disease progression, death, and study termination.
  Defined as patients achieving a complete response [CR] or partial response [PR].

OTHER OUTCOMES:
Tumor markers | Once every 9 weeks (±7 days) from the first day of Envafolimab treatment for a maximum of 2 years until confirmed objective disease progression, death, and study termination.
  The peripheral blood samples of the patients were taken for the determination of tumor-associated Macrophages（TAMs）expression, and the results were analyzed to explore the effect of oxaliplatin on immune remodeling.
Lymphocyte count | Once every 9 weeks (±7 days) from the first day of Envafolimab treatment for a maximum of 2 years until confirmed objective disease progression, death, and study termination.
  Detecting the changes of lymphocyte count to conform the effect of oxaliplatin on tumor immune remodeling.
Adverse events | Envafolimab treatment is performed once per cycle (±7 days), and the last one is completed within 30 days (±3 days) after ending treatment or before starting a new anti-tumor therapy.
  Defined as the incidence of treatment emerge adverse events, treatment related adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Zhengang Yuan, PhD, Principal Investigator — Eastern Hepatobiliary Surgery Hospital, Navy Medical University
Locations (1):
- Easter hepatobiliary surgery hospital, Shanghai, Shanghai Municipality, China